CLINICAL TRIAL: NCT05353738
Title: Evaluation of the Efficacy of Vaccination Against COVID-19 by Screening for Neutralizing Antibodies in Patients Presenting a Neuromuscular Disease With Severe Amyotrophy
Brief Title: Efficacy of Vaccination Against COVID-19 in Patients Presenting a Neuromuscular Disease With Severe Amyotrophy
Acronym: CANNEMUSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/13
Record Dates: First submitted 2022-04-14; First posted 2022-04-29 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Neuromuscular Diseases; COVID-19; Amyotrophy
Keywords: neuromuscular; Amyotrophy; mRNA vaccines; COVID-19; protein neutralization; S infection; vaccine Moderna
MeSH Terms: conditions — Neuromuscular Diseases; COVID-19; Muscular Atrophy | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample at 6 weeks (+/- 4 days) after the second injection of the Moderna vaccine, at 24 weeks (+/- 1 week), at 40 weeks (+/- 1 week) and at 52 or 64weeks (+/- 12 weeks) after the second injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with severe neuromuscular disease: Patient with severe neuromuscular disease and having received vaccination with the Moderna vaccine
  Interventions: Biological: Blood sample for research of anti-xoprs netralizing anti spike; Other: Questionnaire
- Patients groupe témoins négatif: Patient having had a blood sample taken as part of the treatment for virological analysis before anti-COVID 19 vaccination
  Interventions: Biological: Blood sample for research of anti-xoprs netralizing anti spike
- Patients groupe témoins positif: Patient having had a blood sample taken as part of the treatment for virological analysis following infection with the omicron variant.
  Interventions: Biological: Blood sample for research of anti-xoprs netralizing anti spike

INTERVENTIONS:
Biological: Blood sample for research of anti-xoprs netralizing anti spike — The evaluation of the ex vivo efficacy of the Moderna vaccine by the search for anti Spike AcN at 6,24, 40 and 52 or 64 weeks after the second injection of the vaccine.
  The effectiveness of vaccination of CANNEMUSS patients will be evaluated by comparing the antibodies anti-S neutralizers from patients in the CANNEMUSS study to those from patients whose sample was carried out before the pandemic (negative control group) and those of patients infected with the omicron virus (positive control group).
Other: Questionnaire — Evaluation of vaccine efficacy in real life by filling out questionnaires
  Groups: Patients with severe neuromuscular disease

SUMMARY:
Des vaccins sont désormais disponibles en France, dont le vaccin Moderna COVID-19 qui est basé sur la technologie des ARNm. La séquence génétique qu'il contient code pour la protéine Spike (S) de l'enveloppe virale, protéine clé de la pénétration du virus dans les cellules qu'il infecte. Le vaccin ARNm est injecté par voie intramusculaire et pénètre dans les fibres musculaires, qui sont des cellules produisant des protéines en très grande quantité en continu, notamment pour la production de myofibrilles impliquées dans la contraction musculaire. Une fois à l'intérieur de la fibre musculaire, l'ARNm vaccinal est traduit par la machinerie de la fibre musculaire permettant une grande quantité de protéine Spike (S) qui sera présentée au système immunitaire provoquant la réponse vaccinale et notamment les anticorps neutralisants anti-S (NAb). Ces NAb anti-S agissent en perturbant l'interaction entre la protéine S du virus et le récepteur ACE2 (Angiotensin-Converting Enzyme 2), qui sert généralement de " passerelle " entre le virus et la cellule. Une campagne de vaccination est actuellement en cours au MAS-YDK avec le vaccin Moderna. Cette population est donc relativement homogène en termes d'amyotrophie, de non exposition au SARS-CoV-2 et de protocole vaccinal.

DETAILED DESCRIPTION:
COVID-19 is linked to SARS-CoV-2, a new coronavirus that can lead to death. Some neuromuscular patientsare considered at risk for various reasons: cardiomyopathy or rhythm and/or conduction disorder, ventilator insufficiency, severe motor disability with the need for human support for daily activities. Neuromuscular patients with severe amyotrophy are therefore at very high risk of severe forms of COVID-19. A still unpublished study of the French neuromuscular network FILNEMUS showed that in neuromuscular patients the risk of admission to ICU was 21.2% and the lethality rate 9.1%, well above the values observed in the general population. The prevention of COVID-19 is therefore key. Until now, in the MAS-YDK an extremely strict health protocol has been enacted to protect the residents: outings allowed only for medical appointments, 7-day quarantine for any resident returning from outside, routine systematic PCR of patients and caregivers, prohibition of visits by outsiders... This very stringent protocol has been very effective since no resident has presented any symptomatic COVID-19 but this was achieved at the cost of social isolation. Vaccination of both residents and staff is therefore the best avenue of hope for a return to a more normal life. Will vaccines using the muscle cell machinery be effective in amyotrophic patients? Vaccines are now available in France, including the Moderna COVID-19 vaccine which is based on mRNA technology. The genetic sequence it contains encodes the Spike protein (S) of the virus envelope, a protein which is key to the virus's penetration into the cells that it infects. The mRNA vaccine is injected intramuscularly and penetrates muscle fibers, which are cells producing proteins in very large quantities continuously, especially for the production of myofibrils involved in muscle contraction. Once inside the muscle fiber, the vaccine mNRA is translated by the muscle fiber machinery allowing a large amount of Spike protein (S) that will be presented to the immune system causing the vaccine response and in particular anti-S neutralizing antibodies (NAb). These anti-S NAbs work by disrupting the interaction between the virus's S protein and the ACE2 receptor (Angiotensin-Converting Enzyme 2), which usually serves as the "gateway" between the virus and the cell. A vaccination campaign is currently underway at the MAS-YDK with the Moderna vaccine. This population is therefore relatively homogeneous in terms of amyotrophy, lack of exposure to SARS-CoV-2 and vaccine protocol.

ELIGIBILITY:
Inclusion Criteria

- For patients with severe neuromuscular disease:

1. Adult over 18
2. Person with a defined severe neuromuscular pathology by a modified Rankin score ≥ 4
3. Person supported at the YDK pole
4. Person who has received vaccination with the Moderna vaccine, in the quadriceps or deltoid
5. Non-objection of the patient and/or his legal representative to the participation in the study

For patients in the negative control group :

1. Non-objection of the patient to the storage and use in the framework of the CANNEMUSS study of these blood samples from the routine care.
2. Patient having had a blood sample taken as part of the treatment for virological analysis before anti-COVID 19 vaccination.
3. Patient matched in sex and age to a patient included in the study CANNEMUSS.

For patients in the positive control group :

1. Non-objection of the patient to the storage and use in the framework of the CANNEMUSS study of these blood samples from the routine care.
2. Patient having had a blood sample taken as part of the treatment for virological analysis following infection with the omicron variant.

Exclusion Criteria for patients with neuromuscular disease severe

1. Person with symptomatic infection with SARS-CoV-2 proven by a positive PCR
2. Person with Amyotrophic Lateral Sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe neuromuscular disease and patient (groupe temoins) having had a blood sample taken as part of the treatment for virological analysis
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Look for the presence of antibodies anti-Spike neutralizers, 6 weeks after the second injection of the vaccine Moderna against COVID-19 in patients with severe amyotrophy in MAS Yolaine de Kepper. | 6 weeks after the second injection of the Moderna vaccine
  The presence of Ac causing the neutralization of the interaction between the viral protein S and the receptor ACE-2 cells by the syncytia formation inhibition assay.

SECONDARY OUTCOMES:
Confirm the presence of anti-Spike neutralizing antibodies, 6 weeks after the second injection of the Moderna vaccine against COVID-19 by another technique: | 6 week after the second injection of Moderna vaccine
  Neutralization of infection of target cells expressing ACE-2 by a lentivirus expressing protein Sexpressing the protein S
Look for the presence of anti-Spike neutralizing antibodies, 24 weeks after the second injection of the Moderna vaccine against COVID-19 | 24 week after the second injection of the Moderna vaccine against
  Neutralization of the interaction between the viral protein S and the cell receptor ACE-2 by the formation inhibition test of syncytia.
  Neutralization of the infection of target cells expressing ACE-2 by a lentivirus expressing protein S
Look for the presence of neutralizing antibodies to Spike, 52 or 64 weeks after the second injection of the Moderna vaccine against COVID-19 (i.e. approximately 6 months or 9 months after the 3rd dose of reminder) | 52 or 64 week after the second injection of the Moderna vaccine
  Neutralization of the interaction between the viral protein S and the cell receptor ACE-2 by the formation inhibition test of syncytia.
  Neutralization of the infection of target cells expressing ACE-2 by a lentivirus expressing the S protein.
Look for the presence of neutralizing antibodies directed against most recent delta and omicron variants, at all times of study | Throughout study completion, an average 64 week
  Neutralization of the interaction between the viral proteins S delta and omicron and the cellular receptor by inhibition test of variant-adapted syncytia formation
Assessing the effectiveness of vaccination in real life | Throughout study completion, an average 64 week
  - Frequency of COVID-19 cases confirmed by a PCR test or an antigen test that occurred at least 7 days after the second injection of the Moderna vaccine according to the protocol of usual follow-up of SAM YDK
Compare the level of anti-Spike neutralizing antibodies | Throughout study completion, an average 64 week
  Compare the level of anti-Spike neutralizing antibodies of patients with severe disuse atrophy of MAS Yolaine from Kepper to that of a group of patients matched in sex and agewhose sera date from before the pandemic and constitute non-neutralizing negative controls.
Compare the neutralization techniques | Throughout study completion, an average 64 week
  Compare the neutralization techniques developed for MAS YDK patients to some patient sera recently hospitalized with omicron variant infection, such as positive controls for this variant.

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem SOLE, Dr, Principal Investigator — Université Hospital, Bordeaux
Locations (1):
- University Hospital of Bordeaux, Bordeaux, France